CLINICAL TRIAL: NCT06045806
Title: A Randomized, Open-Label, Phase 3 Trial to Compare the Efficacy and Safety of Idecabtagene Vicleucel With Lenalidomide Maintenance Versus Lenalidomide Maintenance Therapy Alone in Adult Participants With Newly Diagnosed Multiple Myeloma Who Have Suboptimal Response After Autologous Stem Cell Transplantation (KarMMa-9)
Brief Title: A Study to Compare the Efficacy and Safety of Idecabtagene Vicleucel With Lenalidomide Maintenance Therapy Versus Lenalidomide Maintenance Therapy Alone in Adult Participants With Newly Diagnosed Multiple Myeloma Who Have Suboptimal Response After Autologous Stem Cell Transplantation
Acronym: KarMMa-9
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Bristol-Myers Squibb (Industry); 2seventy bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA089-1043; 2022-501346-30 (EudraCT Number); U1111-1280-9736 (Other: WHO); NCT06399393 (obsolete NCT alias)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel; Lenalidomide; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: idecabtagene vicleucel; Drug: Lenalidomide; Drug: Fludarabine; Drug: Cyclophosphamide
- Arm B (Active Comparator)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Biological: idecabtagene vicleucel — Specified dose on specified days
  Other Names: BMS-986395; Abecma; bb2121; ide-cel
  Arms: Arm A
Drug: Lenalidomide — Specified dose on specified days
  Other Names: Revlimid; LEN
Drug: Fludarabine — Specified dose on specified days
  Other Names: FLUDARA; BENDARBIN
  Arms: Arm A
Drug: Cyclophosphamide — Specified dose on specified days
  Other Names: ENDOXAN; CYTOXAN
  Arms: Arm A

SUMMARY:
The purpose of this study is to compare the efficacy, safety, and tolerability of ide-cel with lenalidomide (LEN) maintenance to that of LEN maintenance alone in adult participants with Newly Diagnosed Multiple Myeloma (NDMM) who have achieved a suboptimal response post autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria

* Participants aged ≥18 with Newly Diagnosed Multiple Myeloma (NDMM) who has received induction therapy followed by high-dose chemotherapy and autologous stem cell transplantation (ASCT), without subsequent consolidation or maintenance. EXCEPTION: Participant received ≤ 7 days of lenalidomide (LEN) maintenance therapy and the investigator documents that there is no impact to the overall benefit/risk assessment due to the temporary interruption of LEN.
* Participant must have received 4 to 6 cycles of induction therapy, which must contain at a minimum an immunomodulatory drugs (IMiD) and a proteasome inhibitor (PI) (with or without anti-CD38 monoclonal antibody) and must have had a single ASCT 80 to 120 days prior to consent. Note: Participant must not have confirmed progression since commencing induction.
* Participant must have documented response of PR or VGPR at time of consent.
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (participants with ECOG 2 due to pain because of underlying myeloma-associated bone lesions are eligible per investigator's discretion).
* Participant must have recovered to ≤ Grade 1 for any nonhematologic toxicities due to prior treatments, excluding alopecia and Grade 2 neuropathy.

Exclusion Criteria

* Participant with known central nervous system involvement with myeloma.
* Participant has non-secretory MM.
* Participant has systemic and uncontrolled fungal, bacterial, viral, or other infection.
* Participant has history of primary immunodeficiency.
* Participant has previous history of an allogeneic hematopoietic stem cell transplantation or treatment with any gene therapy-based therapeutic for cancer or investigational cellular therapy for cancer or B-cell maturation antigen targeted therapy.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-08-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 50 months after the first participant is randomized
  PFS as assessed by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 60 months after the last participant is randomized
Percentage of Participants with Sustained Minimal Residual Disease Negative (MRDneg) Complete Response (CR) for 12 months | From randomization up to 60 months from randomization
Percentage of Participants with Minimal Residual Disease Negative (MRDneg) Complete Response (CR) | From randomization up to 15 months from randomization
Event-Free Survival (EFS) | Up to approximately 60 months after the last participant is randomized
Duration of Response (DOR) | Up to approximately 60 months after the last participant is randomized
Percentage of Participants with Complete Response (CR) | Up to approximately 60 months after the last participant is randomized
  CR as assessed by IRC
Time to Progression (TTP) | Up to approximately 60 months after the last participant is randomized
  Progression as assessed by IRC
Progression post-next line of treatment (PFS2) | Up to approximately 60 months after the last participant is randomized
Time to Next Treatment (TTNT) | Up to approximately 60 months after the last participant is randomized
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 60 months after the last participant is randomized
Number of Participants Experiencing Adverse Events of Special Interest (AESI) | Up to approximately 60 months after the last participant is randomized
Maximum Observed Plasma Concentration (Cmax) | Up to approximately 60 months after the last participant is randomized
Time of Maximum Observed Plasma Concentration (Tmax) | Up to approximately 60 months after the last participant is randomized
Area Under the Curve (AUC) from time zero to 28 days post infusion (AUC [0- 28D]) | Up to 28 days post infusion
Time of Last Measurable Observed Plasma Concentration (Tlast) | Up to approximately 60 months after the last participant is randomized
Time-to-Definitive Deterioration | Up to approximately 50 months after the first participant is randomized
  Time-to-definitive deterioration based on the European Organization for Research and Treatment of Cancer core quality of life questionnaire EORTC QLQ-C30 global health status/quality of life subscale
Mean Change from Baseline in EORTC QLQ-C30 Selected Subscales | Up to approximately 50 months after the first participant is randomized
  The following subscales on the European Organization for Research and Treatment of Cancer core quality of life questionnaire EORTC QLQ-C30 will be assessed:
  * Global health status/quality of life
  * Physical Functioning
  * Fatigue
  * Pain
Mean Change from Baseline in EORTC QLQ-MY20 Selected Subscales | Up to approximately 50 months after the first participant is randomized
  The following subscales on the European Organization for Research and Treatment of Cancer core quality of life questionnaire EORTC QLQ-MY20 will be assessed:
  * Disease symptoms
  * Side-effects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (100):
- United States (19):
  - Local Institution - 0131, Los Angeles, California
  - Local Institution - 0126, Orange, California
  - Local Institution - 0113, Sacramento, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - Local Institution - 0121, Atlanta, Georgia
  - Local Institution - 0104, Atlanta, Georgia
  - Local Institution - 0151, Boston, Massachusetts
  - Ascension Providence Hospital, Southfield, Michigan
  - M Health Fairview Clinics and Surgery Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Novant Health Cancer Institute - Elizabeth, Charlotte, North Carolina
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Local Institution - 0132, Philadelphia, Pennsylvania
  - Local Institution - 0124, Austin, Texas
  - Local Institution - 0109, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Local Institution - 0007, Camperdown, New South Wales
  - Local Institution - 0005, Brisbane, Queensland
  - Local Institution - 0004, Melbourne, Victoria
  - Local Institution - 0006, Melbourne, Victoria
  - Local Institution - 0008, Melbourne, Victoria
  - Local Institution - 0011, Murdoch, Western Australia
- Austria (2):
  - Local Institution - 0089, Salzburg
  - Local Institution - 0090, Vienna
- Belgium (3):
  - Local Institution - 0083, Anderlecht, Bruxelles-Capitale, Région de
  - Local Institution - 0084, Brussels, Bruxelles-Capitale, Région de
  - Local Institution - 0144, Brussels, Bruxelles-Capitale, Région de
- Canada (3):
  - Local Institution - 0133, Edmonton, Alberta
  - Local Institution - 0001, Hamilton, Ontario
  - Local Institution - 0134, Montreal, Quebec
- Local Institution - 0070, Odense, Region Syddanmark, Denmark
- France (11):
  - Local Institution - 0047, Pessac, Aquitaine
  - Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône
  - Hopital Claude Huriez - CHU de Lille, Lille, Nord
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Pays de la Loire Region
  - Local Institution - 0046, Pierre-Bénite, Rhône
  - Henri Mondor Hospital, Créteil, Val-de-Marne
  - Local Institution - 0028, Villejuif, Val-de-Marne
  - Local Institution - 0029, Poitiers, Vienne
  - Local Institution - 0082, Paris
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse
  - Local Institution - 0031, Paris, Île-de-France Region
- Germany (9):
  - Local Institution - 0072, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0078, Ulm, Baden-Wurttemberg
  - Local Institution - 0077, Nuremberg, Bavaria
  - Local Institution - 0073, Cologne, North Rhine-Westphalia
  - Local Institution - 0087, Leipzig, Saxony
  - Local Institution - 0079, Dresden
  - Local Institution - 0115, Essen
  - Local Institution - 0076, Hamburg
  - Local Institution - 0074, Würzburg
- Greece (4):
  - Local Institution - 0063, Pátrai, Achaḯa
  - Local Institution - 0061, Athens, Attikí
  - Local Institution - 0062, Chaïdári, Attikí
  - Local Institution - 0060, Thessaloniki, Thessaloníki
- Israel (6):
  - Local Institution - 0058, Petah Tikva, Central District
  - Local Institution - 0057, Ramat Gan, Central District
  - Local Institution - 0055, Beersheba, Southern District
  - Local Institution - 0088, Tel Aviv, Tell Abīb
  - Local Institution - 0056, Haifa
  - Local Institution - 0059, Jerusalem
- Italy (3):
  - Local Institution - 0064, Rozzano, Milano
  - Local Institution - 0065, Bologna
  - Local Institution - 0066, Roma
- Japan (10):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiya, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Local Institution - 0085, Isehara, Kanagawa
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Okayama University Hospital, Okayama
  - Local Institution - 0071, Shimotsuke
- Local Institution - 0069, Oslo, Norway
- Poland (6):
  - Local Institution - 0027, Lublin, Lublin Voivodeship
  - Local Institution - 0095, Warsaw, Masovian Voivodeship
  - Local Institution - 0023, Warsaw, Masovian Voivodeship
  - Local Institution - 0022, Gliwice, Silesian Voivodeship
  - Local Institution - 0026, Gdansk
  - Local Institution - 0024, Poznan
- Local Institution - 0091, Bucharest, Romania
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0038, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0043, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Local Institution - 0020, Badalona, Barcelona [Barcelona]
  - Local Institution - 0017, L'Hospitalet Del Llobregat, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0012, Pamplona, Navarre
  - Local Institution - 0021, Madrid
  - Local Institution - 0013, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - Local Institution - 0093, Birmingham, England
  - Local Institution - 0080, London, London, City of
  - Local Institution - 0094, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06045806.html